CLINICAL TRIAL: NCT02276807
Title: RCT of Behavioral Activation for Depression and Suicidality in Primary Care
Brief Title: Improving Mood in Veterans in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 14-047
Record Dates: First submitted 2014-10-08; First posted 2014-10-28 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Depression
Keywords: Depression; Behavioral Symptoms; Mental Disorders; Depressive Disorder; suicidal ideation; primary health care; Veterans
MeSH Terms: conditions — Depression; Behavioral Symptoms; Mental Disorders; Depressive Disorder; Suicidal Ideation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief Behavioral Activation (Experimental): This is a 4-session individual workshop using behavioral activation techniques. Emphasis is placed upon understanding the individuals values and increasing the number of pleasurable activities aligned with the individuals values.
  Interventions: Behavioral: Brief Behavioral Activation
- Usual Care (Active Comparator): This is the usual care condition, where participants often times will be provided with brief treatment in primary care that can take many forms.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Brief Behavioral Activation — This is a 4-session individual workshop using behavioral activation techniques.
  Arms: Brief Behavioral Activation
Other: Usual Care — Primary care patients will be referred to the integrated behavioral health provider to receive brief treatment in primary care.
  Other Names: Usual Care condition
  Arms: Usual Care

SUMMARY:
The purpose of the Improving Mood in Veterans in Primary Care (IIR 14-047) is to evaluate a brief educational individual workshop that is meant to help Veterans better understand feelings of sadness and ways to improve their mood. This study is intended to evaluate and establish the workshop's effectiveness for use with Veterans in primary care settings.

The study involves up to 6 in-person meetings and 6 telephone interviews across a 6-month period of time. Approximately 144 Veterans will participate in the study. Using a procedure like the flip of a coin, the participants will have a one in two chance of receiving the brief educational workshop or treatment as usual condition.

DETAILED DESCRIPTION:
Background:

Depressive symptoms are the most common referral problem to integrated mental health providers within Veteran primary care clinics. Although there exist several empirically-based brief psychotherapies for depression in primary care, the most significant barrier to providing those psychotherapies is treatment duration (e.g., the treatments range from 6-8 sessions of 30-50 minutes) as it does not match typical treatment formats delivered by mental health providers working in primary care (i.e., 1-4 15-30 minute sessions). Therefore, this HSR&D study titled, RCT of Behavioral Activation for Depression and Suicidality in Primary Care, will examine the effectiveness of a brief version of an existing efficacious longer treatment for depression, called behavioral activation.

Objectives:

The overarching objectives of this study are to: 1) examine whether a 4-session manualized behavioral activation intervention (BA-PC) compared to Treatment as Usual (TAU) is effective in reducing self-reported depressive symptoms and subjective secondary outcomes such as sleep impairment and quality of life; 2) examine patient satisfaction, engagement, and receptivity to a 4-session BA-PC; and 3) explore the impact of BA-PC on suicidal ideation.

Methods:

The study will achieve these objectives using a randomized, controlled trial study design that has two conditions (4-session BA-PC and Treatment as Usual). Veterans will be recruited from three VA primary care settings in the Western portion of VISN 2 (Syracuse, Rochester, and Buffalo). The primary inclusion criteria for the study will be a report of depressive symptoms by primary care patients, who are not currently engaged in psychological treatment for depression. A total of 136 Veterans will be targeted for randomization. All Veterans will be assessed every 2 weeks for changes in mood and more comprehensive assessments will be completed at 6, 12, and 24 weeks.

Status:

Recruitment has ended as of 2/26/18 with 140 participants being randomized. Follow-up will continue for another 24 weeks. We are preparing the data for analysis.

ELIGIBILITY:
Inclusion Criteria:

Veterans:

* aged 18 years
* seeking or receiving primary care services at the Syracuse, Canandaigua, or Buffalo VA Medical Centers
* reporting at least moderate depressive symptoms
* stable course of antidepression medications
* stable course of outpatient treatment for anxiety or substance use disorders

Exclusion Criteria:

Veterans who are:

* unable to demonstrate an understanding of the informed consent
* non-English speaking
* reporting imminent risk of suicide
* have an unstable psychiatric condition
* currently involved in treatment for depression
* recently started antidepression medication or outpatient treatment for anxiety or substance use disorder
* currently involved or completed inpatient or intensive outpatient treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Schum Funderburk, PhD, Principal Investigator — Syracuse VA Medical Center, Syracuse, NY
Locations (3):
- United States (3):
  - VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York
  - Canandaigua VA Medical Center, Canandaigua, NY, Canandaigua, New York
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Funderburk JS, Pigeon WR, Shepardson RL, Wade M, Acker J, Fivecoat H, Wray LO, Maisto SA. Treating depressive symptoms among veterans in primary care: A multi-site RCT of brief behavioral activation. J Affect Disord. 2021 Mar 15;283:11-19. doi: 10.1016/j.jad.2021.01.033. Epub 2021 Jan 14. PMID 33516082
- See also: The co-PI's are affiliated with the VA Center for Integrated Healthcare and this website describes current and past research projects similar to the one in this study. — http://www.mirecc.va.gov/cih-visn2/
- See also: Click here for more information about this study: RCT of Behavioral Activation for Depression and Suicidality in Primary Care — http://www.hsrd.research.va.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from three VA primary care clinics in Western New York from March 2015 through March 2018 . Eligible participants (i.e., age > 18 years of age, receiving services in those clinics, and reporting depressive symptoms) were identified via medical record review, study flyers posted in clinics, and direct referrals.
Pre-assignment Details: A two-part screening process identified those eligible to continue into the study based on additional set of eligibility criteria, such as at least moderate symptoms of depression and stable course of antidepressants or outpatient psychotherapy for anxiety, PTSD, or substance use.
Groups:
- Brief Behavioral Activation: This is a 4-session individual workshop using behavioral activation techniques, where content is delivered primarily in the first 2 sessions and 2 additional sessions are used as boosters. Emphasis is placed upon understanding the individuals values and increasing the number of pleasurable activities aligned with the individuals values.
  Brief Behavioral Activation: This is 4-session individual workshop using behavioral activation techniques.
Period: Overall Study
Arm/Group | Brief Behavioral Activation | Usual Care
Started | 68 | 72
12-week Assessment (Participant completed the main outcome measure, but may not have completed all required measures.) | 57 | 63
Completed (Participant completed the main outcome measure, but may not have completed all required measures.) | 50 | 55
Not Completed | 18 | 17
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Lost to Follow-up | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Brief Behavioral Activation: This is a 4-session individual workshop using behavioral activation techniques, where content is delivered primarily in the first 2 sessions and 2 additional sessions are used as boosters. Emphasis is placed upon understanding the individuals values and increasing the number of pleasurable activities aligned with the individuals values.
  Brief Behavioral Activation: This is a 4-session individual workshop using behavioral activation techniques.
- Total: Total of all reporting groups
Arm/Group | Brief Behavioral Activation | Usual Care | Total
Number analyzed (Participants) | 68 | 72 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (14.9) | 54.3 (13.4) | 53.0 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 62 | 66 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 64 | 66 | 130
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 15 | 15 | 30
  White | 43 | 49 | 92
  More than one race | 5 | 6 | 11
  Unknown or Not Reported | 1 | 1 | 2
Patient Health Questionnaire-9 (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The minimum value is 0 and the maximum value is 27. Higher scores mean a worse outcome.
  units on a scale | 16.0 (4.3) | 15.9 (4.5) | 16.0 (4.4)
Beck Scale for Suicidal Ideation (SSI) [Mean (Standard Deviation); unit: units on a scale] — This is focused on the past week's suicidal ideation. The minimum score is 0 and the maximum score is 38. Higher scores mean worse suicidal ideation.
  units on a scale | 2.1 (4.9) | 1.8 (4.1) | 2.0 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Depressive Symptoms at 12 Weeks
Description: The investigators will use the Patient Health Questionnaire-9 (PHQ-9) to assess depressive symptoms at baseline and 12 weeks. The minimum value is 0 and the maximum value is 27. Higher scores mean a worse outcome.
Time Frame: Baseline and 12 weeks
Population: Participants who did not withdraw before week 12 and completed this questionnaire at week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Behavioral Activation | Usual Care
Number analyzed (Participants) | 57 | 63
score on a scale
  PHQ-9 Total Score at Baseline | 15.68 (3.94) | 15.93 (4.38)
  PHQ-9 Total Score at Week 12 | 11.40 (4.94) | 12.56 (5.40)
Statistical Analysis 1: Comparison: Brief Behavioral Activation vs Usual Care; Test type: Superiority; p < 0.05, ANOVA; 2 (Condition: TAU, BA-PC) X 2 (Time: Baseline vs. Week 12) repeated measures ANOVA; Mean Difference (Final Values) = .345

2. Secondary Outcome: Change From Baseline in Quality of Life at 12 Weeks
Description: The investigators will use the Short Form-12 (SF-12) mental health domain to assess quality of life at baseline and 12 weeks. The minimum score is 0 and maximum score is 100. Higher scores mean better quality of life within mental health domain.
Time Frame: Baseline and 12 weeks
Population: Enrolled participants who did not withdraw before 12-weeks and completed this questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Behavioral Activation | Usual Care
Number analyzed (Participants) | 57 | 61
score on a scale
  Total Score at Baseline | 36.18 (15.43) | 34.02 (17.84)
  Total Score at Week 12 | 45.83 (19.53) | 36.68 (19.61)
Statistical Analysis 1: Comparison: Brief Behavioral Activation vs Usual Care; Test type: Superiority; p < 0.05, ANOVA; 2 (Condition: TAU vs. BA-PC) X 2 (time: Baseline vs. week 12) repeated measures ANOVA; Mean Difference (Final Values) = .046

3. Secondary Outcome: Change From Baseline in Sleep Disturbances at 12 Weeks
Description: The investigators will use the Insomnia Severity Index (ISI) to assess sleep disturbances at baseline and 12 weeks. The minimum score is 0 and the maximum score is 28. Higher scores on ISI mean worse sleep.
Time Frame: Baseline and 12 weeks
Population: Enrolled participants who did not withdraw prior to week 12 and completed this assessment measure at week 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Behavioral Activation | Usual Care
Number analyzed (Participants) | 55 | 61
score on a scale
  Total Score at Baseline | 17.07 (7.18) | 16.48 (6.66)
  Total Score at Week 12 | 15.95 (7.48) | 15.77 (6.74)
Statistical Analysis 1: Comparison: Brief Behavioral Activation vs Usual Care; Test type: Superiority; p < 0.05, ANOVA; 2 (Condition: TAU, BA-PC) X 2 (Time: Baseline, Week 12) Repeated Measures ANOVA; Mean Difference (Final Values) = 0.666

4. Secondary Outcome: Change From Baseline in the Level of Reward/Positive Mood When Engaging in Various Experiences at 12 Weeks
Description: The investigators will use the Environmental Observational Reward (EROS) scale to assess level of reward/positive mood at baseline and 12 weeks. The minimum score is 10 and the maximum score is 40. Higher scores mean increased level of positive mood obtained from environment.
Time Frame: Baseline and 12 weeks
Population: Enrolled participants who did not withdraw from the study and completed this assessment measure at week 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Behavioral Activation | Usual Care
Number analyzed (Participants) | 54 | 58
score on a scale
  Total Score at Baseline | 21.91 (3.56) | 20.78 (4.01)
  Total Score at Week 12 | 24.19 (3.93) | 21.17 (4.91)
Statistical Analysis 1: Comparison: Brief Behavioral Activation vs Usual Care; Test type: Superiority; p < 0.05, ANOVA; 2 (Condition: TAU vs. BA-PC) X 2 (Time: Baseline, Week 12) Repeated Measures ANOVA; Mean Difference (Final Values) = 0.014

5. Other Pre Specified Outcome: Change From Baseline in the Level of Intensity of Suicidal Ideation at 12 Weeks
Description: The investigators will use the Beck Scale for Suicidal Ideation to assess intensity of suicidal ideation within the past week at baseline and 12 weeks. The minimum score is 0 and the maximum score is 38. Higher scores mean worse suicidal ideation.
Time Frame: Baseline and 12 weeks
Population: Enrolled patients who did not withdraw from the study and completed this assessment at week 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Behavioral Activation | Usual Care
Number analyzed (Participants) | 57 | 61
score on a scale
  Total Score at Baseline | 2.02 (4.27) | 1.69 (4.13)
  Total Score at Week 12 | 1.19 (3.49) | 1.13 (4.18)
Statistical Analysis 1: Comparison: Brief Behavioral Activation vs Usual Care; Test type: Superiority; p < 0.05, ANOVA; 2 (Condition: TAU vs. BA-PC) X 2 (Time: Baseline vs. Week 12) Repeated Measures ANOVA; Mean Difference (Final Values) = 0.722

ADVERSE EVENTS:
Time Frame: Systematically, serious adverse event data was collected during the medical record review conducted at 12 and 24-week assessments. However, research staff also noted events if participant reported them during brief assessments conducted during the 12-week intervention period.
Arm/Group | Brief Behavioral Activation | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/72
Serious Adverse Events (participants affected / at risk) | 8/68 | 4/72
Other Adverse Events (participants affected / at risk) | 12/68 | 3/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brief Behavioral Activation (N=68) | Usual Care (N=72)
Hospitalization Due to Injury (Injury, poisoning and procedural complications) | 4 (5) | 2 (2)
Hospitalization due to (Surgical and medical procedures) | 1 (2) | 2 (3)
Hospitalization due to Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hospitalization due to Psychiatric Disorders (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brief Behavioral Activation (N=68) | Usual Care (N=72)
Outpatient Surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Clinically Significant Increase in Depressive Symptoms (Psychiatric disorders) | 4 (4) | 1 (1) — Greater than 9 point increase on total score on the PHQ-9
Emergency Room Visit (Injury, poisoning and procedural complications) | 6 (8) | 1 (1)
Distressed Participant Unrelated to Study (Psychiatric disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Limited to a Veteran population willing to engage in a clinical trial, lack of ability to clarify the impact of BA-PC from the impact of BA-PC with regular assessment of depressive symptoms which likely decreased power of sample size unexpectedly

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT02276807/Prot_SAP_000.pdf